CLINICAL TRIAL: NCT04183387
Title: Open-label Randomized Study of Efficacy and Safety of Simvastatin in Uveitis
Brief Title: Simvastatin in Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology (Other)
Responsible Party: Principal Investigator, Ivan Shirinsky, MD, PhD, Head of the Laboratory of Clinical Immunopharmacology, Federal State Budgetary Scientific Institution, Research Institute of Fundamental and Clinical Immunology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMV003
Record Dates: First submitted 2019-11-26; First posted 2019-12-03 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simvastatin and standard treatment (Experimental): 40 mg simvastatin per day for 2 months in addition to conventional treatment of uveitis
  Interventions: Drug: Simvastatin 40mg
- standard treatment (No Intervention): conventional treatment of uveitis

INTERVENTIONS:
Drug: Simvastatin 40mg
  Other Names: simvastatin
  Arms: Simvastatin and standard treatment

SUMMARY:
The study evaluates anti-inflammatory effects and safety of simvastatin in non-infectious uveitis.

DETAILED DESCRIPTION:
3-Hydroxy-3-methyl-glutaryl coenzyme A reductase inhibitors (statins) have been shown to reduce local and systemic inflammation in animal models of various autoimmune disorders including uveitis. In this open-label, randomized study clinical efficacy and tolerability of simvastatin 40 mg/day for 8 weeks is evaluated.

ELIGIBILITY:
Inclusion Criteria:

- diagnosis of active non-infectious uveitis

Exclusion Criteria:

* serious liver or kidney disease
* increased transaminase levels of >1.5 ULN
* planned or active pregnancy
* use of fibrates, nicotinic acid, cyclosporine A, antifungal drugs, macrolide antibiotics, verapamil, and grapefruit juice (>1 L/day).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of corticosteroid sparing control of ocular inflammation | 8 weeks
  Incident cases of corticosteroid sparing control of ocular inflammation will be defined using following criteria:
  1. ≤0.5+ anterior chamber cells, ≤0.5+ vitreous haze, and no active retinal/choroidal lesions; and
  2. ≤10 mg of oral prednisone daily and ≤2 drops of prednisolone acetate 1% (or equivalent) a day;
  The patient should fullfill both criteria to be classified as having corticosteroid sparing control of ocular inflammation

SECONDARY OUTCOMES:
Visual acuity | Baseline, 4 weeks, 8 weeks
  Assessment of visual acuity using the Golovin-Sivtsev table
Anterior chamber cells | Baseline, 4 weeks, 8 weeks
  The grades for anterior chamber cells were 0 (<1 cell), 0.5 (1-5 cells), 1 (6-15 cells), 2 (16-25 cells), 3 (26-50 cells), or 4 (>50 cells)
Anterior chamber flare | Baseline, 4 weeks, 8 weeks
  The grades are the following: 0 (none), 1+ (faint), 2+ (moderate (iris and lens details clear)), 3+ (marked (iris and lens details hazy)), 4+ (intense (fibrin or plastic aqueous)
Vitreous haze | Baseline, 4 weeks, 8 weeks
  Nussenblatt scale:
  0 (no flare), 0.5+ (trace), 1+ (clear optic disc and vessels, hazy nerve fiber layer), 2+ (hazy optic disc and vessels), 3+ (optic disc visible), 4+ (optic disc not visible)
Intraocular pressure | Baseline, 4 weeks, 8 weeks
  Measured using Maklakov tonometer
Changes in tear IL-6 | Baseline, 8 weeks
  Concentrations of IL-6 (pg/ml) in tear samples
Changes in tear IL-8 | Baseline, 8 weeks
  Concentrations of IL-8 (pg/ml) in tear samples
Changes in tear IL-10 | Baseline, 8 weeks
  Concentrations of IL-10 (pg/ml) in tear samples
Changes in tear TNFα | Baseline, 8 weeks
  Concentrations of TNFα (pg/ml) in tear samples
Changes in tear IFN-γ | Baseline, 8 weeks
  Concentrations of IFN-γ (pg/ml) in tear samples
Incidence of corticosteroid sparing control of ocular inflammation | 4 weeks
  Incident cases of corticosteroid sparing control of ocular inflammation will be defined using following criteria:
  1. ≤0.5+ anterior chamber cells, ≤0.5+ vitreous haze, and no active retinal/choroidal lesions; and
  2. ≤10 mg of oral prednisone daily and ≤2 drops of prednisolone acetate 1% (or equivalent) a day;
  The patient should fullfill both criteria to be classified as having corticosteroid sparing control of ocular inflammation

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory of Clinical Immunopharmacology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shirinsky IV, Biryukova AA, Kalinovskaya NY, Shirinsky VS. Tear cytokines as potential biomarkers in non-infectious uveitis: post hoc analysis of a randomised clinical trial. Graefes Arch Clin Exp Ophthalmol. 2020 Aug;258(8):1813-1819. doi: 10.1007/s00417-020-04707-7. Epub 2020 May 6. PMID 32377822